CLINICAL TRIAL: NCT01263444
Title: Efficacy and Safety of Adding the Brinzolamide/Timolol Maleate Fixed Combination (AZARGA®) to Ocular Hypertensive or Glaucoma Patients Uncontrolled on Prostaglandin Monotherapy
Brief Title: Safety and Efficacy of Adding AZARGA® Adjunctive to Prostaglandin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-10-246; 2010-022948-21 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: AZARGA®; Open angle glaucoma; Prostaglandin Therapy
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Glaucoma, Open-Angle | interventions — brinzolamide; Timolol; Azarga; Latanoprost; Travoprost; Bimatoprost; tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azarga (Experimental): Brinzolamide 1% / timolol 0.5% Fixed Combination administered as 1 drop in study eye(s) twice a day (8:00 AM and 8:00 PM) for 12 weeks, at a 5 minute interval from the habitual prostaglandin monotherapy.
  Interventions: Drug: Brinzolamide 1% / timolol 0.5% Fixed Combination; Drug: Habitual prostaglandin monotherapy

INTERVENTIONS:
Drug: Brinzolamide 1% / timolol 0.5% Fixed Combination
  Other Names: AZARGA®
Drug: Habitual prostaglandin monotherapy — Topical ocular therapy used daily as prescribed
  Other Names: Latanoprost; Travoprost; Bimatoprost; Tafluprost

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of adding AZARGA® as a single agent to prostaglandin monotherapy in patients with either ocular hypertension or primary open-angle glaucoma.

DETAILED DESCRIPTION:
This study consisted of 3 study visits (Screening/Baseline, Week 4, and Week 12). Eligible patients self-administered the study medication (AZARGA® Eye Drops), adjunct to their current prostaglandin monotherapy for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, primary open angle (including pigment dispersion) glaucoma in both eyes.
* IOP considered to be safe, in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
* Treated with, and in the Investigator's judgment demonstrated an inadequate response to, prostaglandin monotherapy for a minimum of 4 weeks at Visit 1. Last dose of prostaglandin instilled correctly to put patient within the dosing cycle at Visit 1.
* At Visit 1, have an IOP of ≥ 20 mmHg in at least one eye and ≤ 35 mmHg in both eyes treated with prostaglandin monotherapy.
* Best corrected visual acuity of 1.0 LogMAR or better in each eye.
* In any eye not qualifying as a study eye, IOP should be able to be controlled on no pharmacologic therapy or on prostaglandin monotherapy alone.
* Willing to sign an informed consent form.
* Able to follow instructions and willing and able to attend required study visits.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any component of AZARGA® that is deemed clinically significant in the opinion of the investigator.
* A history of, or at risk for uveitis or cystoid macular edema (CME).
* History of ocular herpes simplex.
* Corneal dystrophies in either eye.
* Concurrent infectious/non infectious conjunctivitis, keratitis or uveitis in either eye (excluding Blepharitis or non-clinically significant conjunctival hyperemia).
* Intraocular conventional surgery or laser surgery in study eye(s) less than 3 months prior to Visit 1.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause apart from glaucoma.
* Use of systemic medications known to affect IOP (e.g. oral beta-adrenergic blockers, alpha-agonists and blockers, angiotensin converting enzyme inhibitors and calcium channel blockers), which have not been on a stable course for 7 days prior to Visit 1 or an anticipated change in the dosage during the course of the study.
* Use of corticosteroids (oral, topical ocular or nasal) within 30 days of Visit 1 and during the course of the study.
* Bronchial asthma or a history of bronchial asthma, bronchial hyper reactivity, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* History of severe allergic rhinitis.
* A condition, which in the opinion of the principal investigator, would interfere with optimal participation in the study, or which would present a special risk to the subject.
* Use of any systemic carbonic anhydrase inhibitors (CAI) (e.g. methazolamide [Neptazane], acetazolamide [Diamox]).
* Severely impared renal function.
* History of an allergy to sulphonamides.
* Bronchial asthma or a history of bronchial asthma, bronchial hyper reactivity, severe allergic rhinitis or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* Pregnant, lactating, or of childbearing potential and not using a reliable method of birth control.
* Any clinically significant, serious, or severe medical condition.
* Participation in any other investigational study within 30 days prior to the screening/baseline visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Durier, Pharm. D, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 study centers located in Austria and 2 study centers located in Spain.
Pre-assignment Details: This reporting group includes all enrolled participants (47).
Period: Overall Study
Arm/Group | Azarga
Started | 47
Completed | 37
Not Completed | 10
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Arm/Group | Azarga
Number analyzed (Participants) | 47
Age, Customized [Number; unit: participants]
  ≤55 Years | 3
  56-65 Years | 10
  66-75 Years | 25
  ≥ 76 Years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Intraocular Pressure (IOP) at Week 12
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement. Only one eye (study eye) contributed to the mean.
Time Frame: Baseline, Week 12
Population: This analysis population includes all patients who received study medication and had at least one on-therapy study visit minus missing responses and/or visit attendance.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azarga
Number analyzed (Participants) | 47
mmHg | -6.0 (3.2)

2. Secondary Outcome: Mean Change From Baseline in IOP Per Prostaglandin Group at Week 12
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement. Only prostaglandin subgroups with ≥ 15 patients were analyzed. Only one eye (study eye) contributed to the mean.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azarga
Number analyzed (Participants) | 47
mmHg
  AZARGA + Latanoprost (n=22) | -7.1 (2.9)
  AZARGA + Travoprost (n=15) | -5.1 (3.4)

3. Secondary Outcome: Mean Change From Baseline in IOP at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azarga
Number analyzed (Participants) | 47
mmHg | -6.0 (3.2)

4. Secondary Outcome: Percentage of Patients Reaching the Target IOP (≤ 18 mmHg)
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). Only one eye (study eye) was assessed.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azarga
Number analyzed (Participants) | 47
percentage of participants | 70.0 [15.9 to 18.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (2 years, 1 month). This analysis group includes all patients who received study medication.
Description: An AE was defined as any untoward medical occurrence in a patient who is administered a study treatment, regardless of causal relationship with the treatment. Reports of AEs were obtained through solicited and spontaneous comments from the patients and through observations by the Investigator as outlined in the study protocol.
Arm/Group | Azarga
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 0/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azarga (N=47)
Pseudo stenocardia (General disorders) | 1

LIMITATIONS AND CAVEATS:
A single-arm, non-randomized study somewhat limits interpretation of efficacy results. A 3-month duration does not allow for long-term safety conclusions; however, data obtained at V2 and V3 did not vary much, indicating a steady state at Month 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.